CLINICAL TRIAL: NCT05095584
Title: Validity of 3 Meter Backward Test in Individuals With Amputations
Brief Title: Validity and Reliability of The 3-Meter Backward Walk Test in Individuals With Lower Limb Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tezel Yıldırım Şahan (Other)
Responsible Party: Sponsor-Investigator, Tezel Yıldırım Şahan, Clinical Researcher, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021/298
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Lower Limb Amputation Knee; Lower Limb Amputation Below Knee (Injury)
Keywords: validity; fall; lower limb amputee; backward walking; reliability
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: crosssectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- validity and reliability of 3 meter backward walking test (Experimental): This study was conducted as "test-retest" design and the psychometric properties of 3-m backward walk test were examined in LLA. The Rivermead Mobility Index, 3-m backward walk test, Berg Balance Scale, Timed Up and Go test were applied to the patients. An experienced physiotherapist performed all these tests. In order to measure test-retest reliability, the second evaluations (retest) were carried out by the same physiotherapist two days following the first evaluation (test). A same evaluator collected data in order to avoid the inter-rater variability error rate between the evaluations. The patient was evaluated at one time of the day for test and retest.
  Interventions: Diagnostic Test: 3 meter backward walk test

INTERVENTIONS:
Diagnostic Test: 3 meter backward walk test — validity and reliability of 3-meter backward walk test in lower limb amputation group

SUMMARY:
Clinicians are routinely required to make decisions about fall risk among lower limb prosthesis users. For these decisions, clinicians should use valid, reliable, quantitative, and multidimensional measures of balance test for individuals with lower-limb amputations. The objective of this study was therefore to establish, validity and reliability for 3 meter backward tests administered to established unilateral lower-limb amputations. This study included a total of 30 lower limb amputees [age (18-65) years]. 3 Meter Backward Walking Test, Rivermead Mobility Index, Timed Up and Go test (TUG) was applied to the patients. The second evaluation (retest) was carried out by the same physiotherapist two days following the first evaluation (test) in order to measure test-retest reliability.

DETAILED DESCRIPTION:
Lower limb amputees (LLA) were recruited from local prosthetic clinics. The inclusion criteria were as follows: unilateral transtibial or transfemoral amputation due to traumatic, dysvascular, or oncologic causes, 18 years of age or older, one or more years of using a prosthesis (i.e., established users), and could walk independently for minimum 10 m). Patients unable to ambulate at least 10 m without an upper extremity assistive device (e.g., cane), have an orthopedic or neurological disease that might influence balance, with complications to their contralateral leg (e.g., joint replacement, arthritis, or wounds), have the severe vision and hearing impairment, amputation of a second limb and individuals with stump wounds and gait problems were not enrolled in the research. This study was conducted as a "test-retest" design and the psychometric properties of the 3-m backward walk test were examined in LLA. The Rivermead Mobility Index, 3-m backward walk test, Berg Balance Scale, Timed Up, and Go test was applied to the patients. An experienced physiotherapist performed all these tests. In order to measure test-retest reliability, the second evaluations (retest) were carried out by the same physiotherapist two days following the first evaluation (test). The same evaluator collected data in order to avoid the inter-rater variability error rate between the evaluations. The patient was evaluated at one time of the day for test and retest.

Participants were asked to walk backward within the 3-meter distance marked with black bands on the floor. Participants were asked to walk backward as soon as possible with the "walk" command, to stop at the end of 3 meters, and the elapsed time was recorded in seconds.

Individuals were allowed to look back if they wanted to. To prevent the individual from falling during walking backward and to support the individual, the physiotherapist who made the evaluation walked with an amputee. Measurements were made 3 times and the average time was recorded. During walking backward, there is a greater feeling of insecurity compared to walking forward and causes fear of falling. Therefore, the therapist stood approximately half a meter behind the patient during the test.

ELIGIBILITY:
Inclusion Criteria:

* unilateral transtibial or transfemoral amputation due to traumatic, dysvascular, or oncologic causes,
* 18 years of age or older,
* one or more years of using a prosthesis (i.e., established users),
* could walk independently for a minimum of 10 m).

Exclusion Criteria:

* ambulate at least 10 m without an upper extremity assistive device (e.g., cane),
* have an orthopedic or neurological disease that might influence balance,
* with complications to their contralateral leg (e.g., joint replacement, arthritis, or wounds),
* have severe vision and hearing impairment,
* amputation of a second limb and individuals with stump wounds and gait problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
validity and reliability of 3 meter backward walking test in lower limb amputees | 4 weeks
  validity and reliability

CONTACTS AND LOCATIONS:
Locations (1):
- Tezel Yıldırım Şahan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abit Kocaman A, Aydogan Arslan S, Ugurlu K, Katirci Kirmaci ZI, Keskin ED. Validity and Reliability of The 3-Meter Backward Walk Test in Individuals with Stroke. J Stroke Cerebrovasc Dis. 2021 Jan;30(1):105462. doi: 10.1016/j.jstrokecerebrovasdis.2020.105462. Epub 2020 Nov 13. PMID 33197801